CLINICAL TRIAL: NCT06030908
Title: Functional Outcomes and Return to Sports After Surgical Treatment of Insertional Achilles Tendinopathy With Tendon Debridement and Anchor Refixation.
Brief Title: Outcome After Surgical Reconstruction of the Achilles Tendon Insertion.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Krankenhaus Barmherzige Schwestern Linz (Other)
Responsible Party: Sponsor
Other Study IDs: AST_2023
Record Dates: First submitted 2023-08-28; First posted 2023-09-11 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Achilles Tendinopathy; Insertional Achilles Tendinopathy
Keywords: insertional; Achilles Tendinopathy; surgery; sport

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study Population: Patients who underwent surgical reconstruction of the Achilles tendon insertion using a knotless, double-row anchor system.
  Interventions: Procedure: Reconstruction of Achilles tendon insertion

INTERVENTIONS:
Procedure: Reconstruction of Achilles tendon insertion — knotless double-row anchor fixation of the achilles tendon insertion

SUMMARY:
The purpose of this study is to evaluate the functional outcomes and sports ability after surgical treatment of insertional Achilles tendon tendinopathy using tendon detachment, debridement, and double-row anchor refixation.

DETAILED DESCRIPTION:
The lifetime risk of Achilles tendon pain is approximately 6%, one-third of whom complain of pain at the bony attachment of the Achilles tendon to the calcaneus.

Primary treatment of these insertional tendinopathies is always nonsurgical with physical therapy, orthotics, shock wave therapy, or various forms of injections. If there is no response to therapy, surgery is warranted after three to six months. In this procedure, the tendon is detached from the bone, the damaged portions of the tendon are removed, bony prominences are rounded, and finally the tendon attachment is reconstructed and fixed with anchors. Various anchor systems are available for this purpose.

The double-row anchor system used by the investigators in recent years allows stable, knotless, two-dimensional refixation of the Achilles tendon to the calcaneus and thus permits rapid rehabilitation. Recent studies show good functional results 33 months after reconstruction of the Achilles tendon attachment with the "Speed Bridge" System. To the best of our knowledge, however, there are no studies to date on sports ability after this operation.

The investigators are therefore conducting a retrospective collection of clinical patient data combined with a planned (prospective) questionnaire survey of patients with insertional Achilles tendon tendinopathy who received surgical treatment with tendon refixation.

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent reconstruction and double-row anchor refixation of the Achilles tendon insertion due to an insertional tendinopathy of the Achilles tendon.

Exclusion Criteria:

* Lack of informed consent
* Revision surgery
* Patients who had another operation on the same leg during the same procedure or 6 months later

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients who underwent reconstruction and double-row anchor refixation of the Achilles tendon insertion between 01/2018 and 10/2021.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Return to sports Rate | minimum 12 months from surgery to follow-up
  in percentage compared to preoperatively

SECONDARY OUTCOMES:
Number of sport units per week, sport disciplines practiced | minimum 12 months from surgery to follow-up
  in absolute numbers
Length of sport units | minimum 12 months from surgery to follow-up
  in minutes
Range of motion after surgery | minimum 12 months from surgery to follow-up
  in degrees
Subjective change of instability after surgery | minimum 12 months from surgery to follow-up
  Visual analog scale; 0-10; 0 means no instability, 10 means worst instability
Change of pain after surgery | minimum 12 months from surgery to follow-up
  Visual analog scale; 0-10; 0 means no pain, 10 means worst pain
Satisfaction with result | minimum 12 months from surgery to follow-up
  Visual analog scale; 0-10; 0 means not satisfied, 10 means maximum satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Ordensklinikum Linz, Barmherzige Schwestern Abteilung Orthopädie, Linz, Austria